CLINICAL TRIAL: NCT05521009
Title: Comparison of Adhesive and Non-adhesive Endotracheal Tube Holder Applied in Intensive Care in Terms of Bacterial Colonization
Brief Title: Comparison of Adhesive and Non-adhesive Endotracheal Tube Holder Applied
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Zuhal Gülsoy, Director, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CU
Record Dates: First submitted 2022-08-24; First posted 2022-08-30 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Infection; Intensive Care; Nurses Role; Patient Care
Keywords: intensive care; endotracheal tüp; endotracheal tube fixation; infektion; nursing care
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endotracheal tube fixation (Experimental): Tube fixation will be performed using a bandage in one of the groups. The patients identified with the bandage will form the control group of the study. The group of the patients to be included in the groups will be determined by drawing lots. Except for the different fixation material, no different application will be made to the patients in oral care. As soon as the patients are intubated, a swab will be taken twice, from the outer surface of the endotracheal tube from the fixation distance, and from the same area 3 days after intubation
  Interventions: Other: Control grup, sticky tube holder
- Enfection (Experimental): Tube fixation will be performed with adhesive tube fixation material to one of the groups. In which group the patients to be included in the groups will be will be determined by drawing lots. Except for the different fixation material, no different application will be made to the patients in oral care. As soon as the patients are intubated, a swab will be taken twice, from the outer surface of the endotracheal tube from the fixation distance, and from the same area 3 days after intubation.
  Interventions: Other: Control grup, sticky tube holder

INTERVENTIONS:
Other: Control grup, sticky tube holder — In patients using adhesive tube holders and non-adhesive tube holders, it will be investigated whether there is bacterial growth on the tube.
  Other Names: adhesive tube holder

SUMMARY:
Mechanical ventilation is the continuation of respiratory function from outside by means of special devices until adequate oxygenation is provided by the patient's own respiratory functions in patients whose oxygenation is not sufficient for any reason. . Mechanical ventilation support is provided to patients with respiratory distress with a medical device called an endotracheal tube (ET) inserted through the mouth or nose. Endotracheal intubation is the most common access route for invasive mechanical ventilation (MV) in critical care areas such as the intensive care unit. As in the intensive care unit, as the tube insertion time increases, it becomes very important to fix the tube so that it does not come out. One of the most important and most common complications after ET placement is unplanned extubation. Correct tube detection is the best way to prevent unplanned extubation. In current clinical practice, there are several methods for securing ETs, including adhesive or cloth tapes and endotracheal tube attachment devices. Although there are many types of endotracheal tube holders today, the use of bandages or tapes is still the most commonly used method. Different endotracheal tube fixation techniques used have different advantages and complications. Skin injury and allergy due to adhesive tapes, which are frequently used in the detection of ET, are complications that can be seen in every patient and age group. Endotracheal tube fixation methods may increase the risk of infection due to the material from which they are produced.We planned this study to determine whether the endotracheal tube fixation tie or the gauze fixation from my tube fixation materials contains pathogens, and if so, the pathogen hosting rates.

DETAILED DESCRIPTION:
Mechanical ventilation is the continuation of respiratory function from outside by means of special devices until adequate oxygenation is provided by the patient's own respiratory functions in patients whose oxygenation is not sufficient for any reason. Today, mechanical ventilation is used for various purposes in different environments such as the operating room, intensive care, emergency room and home. Mechanical ventilation support is provided to patients with respiratory distress with a medical device called an endotracheal tube (ET) inserted through the mouth or nose. Endotracheal intubation is the most common access route for invasive mechanical ventilation (MV) in critical care areas such as the intensive care unit. Laryngeal trauma, bronchospasm, hypotension, hypoxemia, airway perforation, and vertebral trauma during endotracheal intubation. many potential complications such as colon injury can be seen. As in the intensive care unit, as the tube insertion time increases, it becomes very important to fix the tube so that it does not dislodge. One of the most important and most common complications after ET placement is unplanned extubation. Correct tube detection is the best way to prevent unplanned extubation. In current clinical practice, there are several methods for securing ETs, including adhesive or cloth tapes and endotracheal tube attachment devices. Although there are many types of endotracheal tube holders today, the use of bandages or tapes remains the most commonly used method. Poor detection of ET may lead to misalignment, slippage, trauma to the airways, or accidental extubation. Excessive pressure of ET detection on facial tissue may cause permanent skin and mucosal damage. Different endotracheal tube fixation techniques used have different advantages and complications. Skin injury and allergy due to adhesive tapes, which are frequently used in the detection of ET, are complications that can be seen in every patient and age group.

There are studies in the literature showing that endotracheal tube fixation methods may increase the risk of infection in relation to the material from which they are produced. In the literature review, it is stated that as a result of the contamination of the adhesive tape with oral secretions in the detection of ET, it prepares an environment for the proliferation of pathogenic microorganisms and increases the risk of infection. ET adhesive tapes cover the mouth in a way that makes oral hygiene difficult due to its wide width. From time to time, the sticky part is left open, which creates an environment prone to infection as a result of the adhesion of unwanted substances such as infection and hair. The evidence is that pathogens are present on existing adhesive tape, and many researchers have found that the adhesive tape is contaminated outside of its original packaging. On the other hand, cotton tapes when tied horizontally (traditionally) cause increased secretions to be absorbed and may therefore harbor infection.

There are currently 3 tube fixation materials in of researches hospital. The first of these is fixation with a sticking tape, the second is fixation with gauze, and the third is commercial cotton tube ties. The sticking tape is not preferred for long-term tube fixation, since its stickiness is lost by getting wet due to the secretion in the mouth of the patients in the intensive care unit. Fixation with gauze is more time consuming in terms of use and requires the use of a cutting tool such as a scalpel to cut the lace, and it is not preferred because it may cause damage and injuries to the tube. Commercial fastening ties, which are easier to use but have adhesive tape at the contact point with the tube, are used in the institution. The pathogen harboring risk that applies to adhesive tapes may also apply to these fixing materials. In addition, as the cares get dirty, the tube fixation material is changed by the nurses and oral care is provided. Each time the fixings are opened, some adhesive tape remains on the tube and a rough surface forms on the tube over time. It is known that pathogen hosting rates are high on rough floors. Choosing the appropriate fixation material in terms of patient safety and performing their care correctly are among the important responsibilities of the intensive care nurse. This study was planned to compare the pathogen harboring rates of endotracheal tube fixation tie and gauze fixation, which are tube fixation materials.

ELIGIBILITY:
Inclusion Criteria:

Patients over 18 years of age, Patients connected to MV, with endotracheal tube, Patients without intraoral damage patients Patients staying with the tube for three days

Exclusion Criteria:

Patients whose tube is removed, Patients who died without a second microbiological swab sample Patients who changed without a second microbiological swab sample

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
physiological parameter | 6 mounts
  After endotracheal intubation, the level of the tube must be maintained so that the tube does not become dislodged. If the tube enters the lungs too much or goes out, it prevents the patient from breathing. For this reason, it will be recorded that the tube stops at the distance it is inserted.

SECONDARY OUTCOMES:
physiological parameter | 6 mounts
  Pathogen formation associated with fixation material around the endotracheal tube may increase the patient's risk of developing ventilator-associated pneumonia. The presence of potential and the amount of pathogen will be determined by microbiological examination of the tube fixation material area.

CONTACTS AND LOCATIONS:
Overall Officials: zuhal gulsoy, Principal Investigator — Nurse
Locations (1):
- Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harris PN, Ashhurst-Smith C, Berenger SJ, Shoobert A, Ferguson JK. Adhesive tape in the health care setting: another high-risk fomite? Med J Aust. 2012 Jan 16;196(1):34. doi: 10.5694/mja11.11211. No abstract available. PMID 22256926
- [Background] Landsperger JS, Byram JM, Lloyd BD, Rice TW; Pragmatic Critical Care Research Group. The effect of adhesive tape versus endotracheal tube fastener in critically ill adults: the endotracheal tube securement (ETTS) randomized controlled trial. Crit Care. 2019 May 7;23(1):161. doi: 10.1186/s13054-019-2440-7. PMID 31064406
- See also: Related Info — http://www.apsf.org/newsletters/html/2011/winter/10_ivtape.htm